CLINICAL TRIAL: NCT01229345
Title: The Interactive Effect of Breakfast Consumption and Exercise on Metabolism, Appetite and Cognitive Function
Brief Title: Effect of Exercise With or Without Breakfast, on Metabolism, Appetite and Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, Javier Gonzalez, PhD Student, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 32W3
Record Dates: First submitted 2010-10-12; First posted 2010-10-27 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: Energy Balance,; Appetite,; Cognitive Function.
MeSH Terms: interventions — Breakfast; Exercise

ARMS (4):
- Breakfast & exercise (Experimental)
  Interventions: Drug: Breakfast & exercise
- Breakfast & no exercise (Experimental)
  Interventions: Drug: Breakfast & exercise
- No breakfast & exercise (Experimental)
  Interventions: Drug: Breakfast & exercise
- No breakfast & no exercise (No Intervention)

INTERVENTIONS:
Drug: Breakfast & exercise — 1859 kJ breakfast vs fast, exercise at 60% maximum aerobic capacity to expend 1859 kJ.
  Arms: Breakfast & exercise; Breakfast & no exercise; No breakfast & exercise

SUMMARY:
The purpose of this study is to assess the effect of eating breakfast in combination with exercise on fat usage, appetite and brain performance later in the day.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged 18-45 years
* BMI 18.5-24.9 kg/m2
* Physically active: able to run for 1 h at a moderate pace
* Healthy

Exclusion Criteria:

* Smokers
* Food allergies
* Metabolic disorders
* Restrained eaters (equivalent of >7 for restrained on TFEQ)
* Consuming herbal/dietary supplements
* History of head trauma
* Learning difficulties
* ADHD
* Dyslexia
* History of migraines
* Gastric problems

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Energy balance | 24 h
  Energy balance (kJ/kcal) will be assessed by an ad libitum test meal provided at 5 h minus energy expenditure estimated by indirect calorimetry.

SECONDARY OUTCOMES:
Blood glucose | 1.5 h area under the curve, post-consumption of a liquid snack
Serum insulin | 1.5 h area under the curve, post-consumption of a liquid snack
Subjective appetite ratings | 1.5 h area under the curve, post-consumption of a liquid snack and following an ad libitum test meal
  Participants will be asked to complete visual analogue scales (VAS).
Cognitive function measurements | 1.5 h area under the curve, post-consumption of a liquid snack and following an ad libitum test meal
  Reaction time, short-term memory, speed of processing, attention.
Mood | 1.5 h area under the curve, post-consumption of a liquid snack and following an ad libitum test meal
  Participants will be asked to complete visual analogue scales (VAS).
Energy expenditure | 1.5 h mean following a liquid snack
  Measured by indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Emma J Stevenson, PhD, Principal Investigator — Northumbria University
Locations (1):
- Brain, Performance and Nutrition Centre, Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom